CLINICAL TRIAL: NCT00563238
Title: Use of Prophylactic Beta Blockade to Prevent Peri-extubation Cardiac Ischemia and Congestive Heart Failure
Brief Title: Beta-blocker Before Extubation
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Gregory A. Schmidt (Other)
Responsible Party: Sponsor-Investigator, Gregory A. Schmidt, Professor, University of Iowa
Organization: University of Iowa (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 200708711
Record Dates: First submitted 2007-11-21; First posted 2007-11-26 (Estimated); Last update posted 2017-02-28 (Actual); Status verified 2017-02

CONDITIONS: Myocardial Ischemia
Keywords: Extubation
MeSH Terms: conditions — Myocardial Ischemia | interventions — Metoprolol

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention)
- Metoprolol (Active Comparator)
  Interventions: Drug: Metoprolol

INTERVENTIONS:
Drug: Metoprolol — Metoprolol administered intravenously in 2.5mg boluses until the resting heart rate falls by 10% from baseline to a maximum dose of 10mg, or until there is any apparent adverse reaction.
  Arms: Metoprolol

SUMMARY:
Silent myocardial ischemia is known to occur in the general medical intensive care unit population immediately following tracheal extubation. We believe these patients are at risk for primary cardiac events in the 4 hours immediately following extubation. Metoprolol is a selective beta-1 antagonist, with little to no beta-2 activity at low and moderate doses. The cardioprotective effects of beta blockade have been well documented in randomized controlled trials. In patients undergoing extubation, prophylactic use of intravenous metoprolol may reduce post-extubation ischemia events as well as precursors of cardiogenic pulmonary edema (atrial and ventricular wall tension). Our primary hypothesis is that prophylactic metoprolol (titrated to reduce resting heart rate by at least 10%) prior to tracheal extubation will reduce the rate of ischemia as judged by ST segment analysis.

ELIGIBILITY:
Inclusion Criteria:

* Adult medical or cardiac intensive care unit patients on mechanical ventilation who have known coronary artery disease or have at least 2 of the following risk factors for coronary artery disease:

  * Cigarette smoking
  * Hypertension (BP 140/90 or antihypertensive medication)
  * Low HDL-cholesterol (HDL-C) (<40 mg/dL [1.03 mmol/L])
  * Family history of premature CHD (in male first degree relatives <55 years, in female first degree relative <65 years)
  * Age (men 45 years, women 55 years)
  * Diabetes mellitus
  * Symptomatic carotid artery disease
  * Peripheral arterial disease
  * Abdominal aortic aneurysm

Exclusion Criteria:

* Arterial hypotension, defined as mean arterial pressure < 60 mmHg or requiring any intravenous vasoactive medication.
* The presence of known reactive airway disease.
* Resting heart rate of <60 in the period prior to tracheal extubation..
* The presence of decompensated congestive heart failure, defined as requiring continuous infusion of an inotropic agent.
* Known hypersensitivity to beta-blockers or any other contraindication to their use.
* Subjects younger than 18 years of age.
* Inability to obtain consent from the subject or the subjects authorized representative.
* Pregnancy
* Digoxin therapy
* Current therapy with a beta-blocker

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2007-11; Primary Completion 2009-12 (Estimated); Study Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
The rate of ischemia as judged by ST segment analysis in the 4h following extubation | 4 hours

SECONDARY OUTCOMES:
Rate-pressure product following extubation | 30min, 2h, 4h
Troponin T elevations, the incidence of cardiogenic edema, and the rate of reintubation | 48h
Pro-BNP levels | 30min

CONTACTS AND LOCATIONS:
Overall Officials: Gregory A Schmidt, MD, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa Hospitals and Clinics, Iowa City, Iowa, United States